CLINICAL TRIAL: NCT06674213
Title: Comparison of Ilioinguinal/Iliohypogastric Nerve Block, Erector Spine Nerve Block and Retrolaminar Nerve Block in Terms of Post-operative Pain in Inguinal Hernia Operations
Brief Title: Comparison of Three Nerve Blocks in Terms of Post-operative Pain in Inguinal Hernia Operations
Status: Completed | Type: Observational
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, DİDEM ONK, Professor Dr., Erzincan University
Other Study IDs: ErzincanU-ANESTEZİ-DO-01
Record Dates: First submitted 2024-10-14; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain
Keywords: Pain, Postoperative; Hernia, Inguinal; erector spinae plane block; retrolaminar block; Ilioinguinal/iliohypogastric nerve
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Grup I-İlioinguinal/İliohipogastrik Nerve Block: Ilioinguinal/Iliohypogastric nerve block will be applied under ultrasound guidance. Pain measurements were evaluated 24 hours after surgery. Pain measurement will be evaluated according to the VAS scale.
- Grup II-Erektör Spine Nerve Block: Erector spine plane block will be applied under ultrasound guidance. Pain measurements were evaluated 24 hours after surgery. Pain measurement will be evaluated according to the VAS scale.
- Grup III-Retrolaminer Nerve Block: Retrolaminar block will be applied under ultrasound guidance. Pain measurements were evaluated 24 hours after surgery. Pain measurement will be evaluated according to the VAS scale.

SUMMARY:
The purpose of this study is to compare the postoperative pain of patients who underwent Inguinal Hernia surgery and the differences between 3 different postoperative nerve block techniques on postoperative pain. It will be investigated which block has the higher effect on postoperative pain and can be used to control the patient's pain.

DETAILED DESCRIPTION:
This observational clinical study was conducted on the General Surgery operating table in Erzincan Mengücek Gazi Training and Research Hospital operating room between 3 April and 3 October 2023, after receiving approval from Erzincan Binali Yıldırım University Faculty of Medicine Ethics Committee dated 30.03.2023 and decision number 2023-07/8. Patients planned to be included in the study were included in the study after they were informed about the study and their consent was obtained.

Criteria for inclusion in the study:

* Having ASA 1 and 2 risk scores
* Primary unilateral Inguinal Hernia operation was performed
* Patients between the ages of 18-60

Exclusion criteria:

* Patients with ASA risk score of 3 and above
* Patients who underwent Recurrent Inguinal Hernia operation
* Patients who underwent Bilateral Inguinal Hernia operation
* Pregnant Patients
* Those with Neuromuscular Disease
* Patients with Uncontrolled Diabetes Mellitus
* Patients who do not accept the study
* Patients with Cognitive Dysfunction
* Patients with a history of Local Anesthetic Drug Toxicity
* Patients with a History of Cerebrovascular Disease
* Patients with Neurological Dysfunction
* Patients with Bleeding Diathesis
* Patients with spinal deformity

Power analysis was performed by examining sample articles. As the sample size: When Type 1 error (α) = 0.005 and power (1-β) = 0.80 were selected, 3 groups (Group 1: Ilioinguinal-iliohypogastric nerve block; Group 2: Erector spine nerve block; Group 3: Retrolaminar nerve block) In this study, postoperative pain scores will be compared; When the effect size (Cohen -f) = 0.25 was taken, a total of 159 people were included in the study, 53 people in each group, according to one-way analysis of variance. However, since our study was a follow-up study, a total of 174 people were included in the study with a loss prediction of 10%, taking into account the losses. Data analysis was done in IBM SPSS 25.0 (SPSS Inc., Chicago, IL, USA) package program.

After the patients were taken to the operating table, standard ASA monitoring (electrocardiogram, non-invasive blood pressure, O2 saturation, body temperature) was applied. All patients underwent spinal anesthesia. 174 patients between the ages of 18-60, with ASA I-II, were included in the study after the surgical procedure was completed after anesthesia application. The demographic characteristics of the patients to be included in each group were shown to be similar and they were included in the group. Esaote MyLab™ Six was used as USG in all blocks. In Group I patients, under USG guidance, a high-frequency linear USG probe was placed on the imaginary line connecting the SIAS (spina iliaca anterior superior) and umbilicus in the supine position. The ilioinguinal/iliohypogastric nerves were scanned with USG until they were seen in the fascia between the internal oblique muscle and the transversus abdominis muscle. Visualization of the Circumflex Iliac Artery in the intermuscular fascia was considered as another anatomical landmark to confirm that we were in the correct injection plane. After the injection site was determined, the block needle was entered into the USG in plane at an angle of approximately 30-45 degrees in the craniocaudal direction, it was confirmed that it was not in the intravenous area with negative pressure, and local anesthetic was injected and its spread was monitored. In the Lumbar region ESPB, the high-frequency linear probe was placed parasagittally 3-5 cm lateral to the median line (spinous processes) in Group II patients in the prone position under USG guidance to visualize the transverse processes. After the transverse protrusion was seen, the needle was entered into the skin by giving the probe an angle of approximately 30-45 degrees in the craniocaudal direction. The application site was determined as the fascia between the erector spinae muscle and the transverse process. In-plane technique, after the needle touched the posterior end edge of the transverse process, it was confirmed that it was not in the intravenous area with negative pressure. Then, its distribution was visualized with ultrasonography (USG). The procedure was completed by observing the local anesthetic distribution in the craniocaudal direction. After visualizing the spinous processes in the lumbar region with a high-frequency linear probe in the prone position of Group III patients under USG guidance, the probe was advanced 1-2 cm laterally and the laminae were visualized in the parasagittal plane. After the retrolaminar region was determined, the block needle was entered into the USG in plane, at an angle of approximately 30-45 degrees in the craniocaudal direction. After contacting the lamina and confirming that it was not in the intravenous area with negative pressure, local anesthetic was injected and its spread was monitored. Pain scores were evaluated with a 10-scale VAS scale (0: No pain; 10: The most severe pain) at 0, 4, 12, and 24 hours after surgery. In the postoperative period, the need for additional analgesics, VAS values and other complications were recorded. Data were obtained from anesthesia records and patients were followed with a data tracking form from the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Having ASA 1 and 2 risk scores
* Primary unilateral Inguinal Hernia operation was performed
* Patients between the ages of 18-60

Exclusion Criteria:

* Patients with ASA risk score of 3 and above
* Patients who underwent Recurrent Inguinal Hernia operation
* Patients who underwent Bilateral Inguinal Hernia surgery
* Pregnant Patients
* Those with Neuromuscular Disease
* Patients with Uncontrolled Diabetes Mellitus
* Patients who do not accept the study
* Patients with Cognitive Dysfunction
* Patients with a history of Local Anesthetic Drug Toxicity
* Patients with a History of Cerebrovascular Disease
* Patients with Neurological Dysfunction
* Patients with Bleeding Diathesis
* Patients with spinal deformity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 159 patients will be included in the study. However, since our study is a follow-up study, a total of 174 patients will be included in the study with a loss prediction of 10%, taking into account the losses. Patients will between the ages of 18-60, who are planned for elective unilateral inguinal hernia surgery by the General Surgery clinic, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 24 Hours
  The patient's Pain Score (VAS Scale) will be evaluated at the 0th hour, 4th hour, 12th hour and 24th hour postoperatively. VAS scale; 0: no pain, 10: very severe, unbearable pain. For postoperative patient monitoring, a physician who does not know the type of block applied will evaluate the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Unıversitesi, Erzincan, Merkez, Turkey (Türkiye)